CLINICAL TRIAL: NCT00170443
Title: A Phase II Evaluation of the Reactogenicity and Immunogenicity of Different Doses of Intramuscular Trivalent Baculovirus-expressed Influenza HA Vaccine in Healthy Elderly Adults
Brief Title: Trivalent rHA Dose Escalation Study in Elderly Subjects
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Robert Johnson, HHS/NIAID/DMID
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 03-119
Record Dates: First submitted 2005-09-09; First posted 2005-09-15 (Estimated); Last update posted 2011-08-12 (Estimated); Status verified 2006-04

CONDITIONS: Influenza
Keywords: Influenza, Baculovirus, Immunogenicity, Geriatrics
MeSH Terms: conditions — Influenza, Human

INTERVENTIONS:
Biological: rHAO Trivalent Influenza Vaccine

SUMMARY:
This study will compare the safety and immunogenicity of three different dose levels of an experimental recombinant influenza HA protein vaccine to a standard inactivated influenza vaccine in heallthy elderly subjects ages 65-80. Blood and nasal secretions for assessment of antibody responses will be obtained from all subjects prior to and one month after vaccination.

DETAILED DESCRIPTION:
Approximately 400 healthy, ambulatory adults ages 65-80 will be randomized into one of four study groups to receive a single immunization of a licensed trivalent inactivated influenza vaccine or one of three dose levels of an investigatioanl trivalent recombinant influenza HA protein vaccine. The study will be conducted in 2 stages. In the first stage, 80 subjects will be randomized (20 per group) and receive one vaccination on Day 0. Safety will be evaluated after Stage 1 subjects have completed a 7 day follow-up. Enrollment of Stage 2 subjects will begin after the safety data for Stage 1 has been reviewed. In Stage 2, 320 subjects will be randomized (80 per group) and receive one vaccination on Day 0. Blood and nasal secretions will be collected prior to an approximately one month after vaccination to assess antibody responses.

ELIGIBILITY:
Inclusion Criteria:

* Medically stable adult age 65 -80.
* Able to give informed consent.
* Able to comply with all study procedures.
* Community dwelling.

Exclusion Criteria:

* History of immunodeficiency or treatment with immunosuppressive medications. (use of inhaled steroids or of topical steroids is not considered immunosuppressive).
* Allergy to eggs, egg proteins, thimerosal, or other vaccine components.
* Acute febrile illness or upper respiratory tract illness within 72 hours of vaccination.
* Life expectancy less than 6 months.
* Use of experimental vaccines or medications within one month of study entry.
* Receipt of parenteral immunoglobulin within one month of study entry.
* Any acute or chronic condition which in the opinion of the investigator would render vaccination unsafe or interfere with the evaluation of response.

Ages: 65 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 399 (Actual)
Dates: Study Completion 2004-06

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - University of Rochester, Rochester, New York
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Baylor College of Medicine, Houston, Texas